CLINICAL TRIAL: NCT06067958
Title: Intranasal Dexmedetomidine for Pain Management During Screening for Retinopathy of Prematurity: a Crossover Randomized Controlled Trial
Brief Title: Intranasal Dexmedetomidine for Pain Management During Screening for Retinopathy of Prematurity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Sagee Nissimov, Principal Investigator, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0096-23-ASF
Record Dates: First submitted 2023-09-12; First posted 2023-10-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Retinopathy of Prematurity; Dexmedetomidine
Keywords: Retinopathy of Prematurity; Dexmedetomidine; Pain; Analgesia; Premature Infant Pain Profile - Revised
MeSH Terms: conditions — Retinopathy of Prematurity; Pain; Agnosia | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This will be a crossover, prospective randomized controlled trial. Block randomization will be performed before the first eye examination. Every participant will undergo two eye examinations - one following exposure to dexmedetomidine and one following placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The units pharmacologist will be responsible for patient assignment and preparation of the medication / placebo syringes but will remain blinded to the other aspects of the trial. The patient's nurse, attending physician, ophthalmologist, investigator and outcome assessor will remain blinded to the patient allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Intranasal Dexmedetomidine 2 microgram/kilogram, 30 minutes before eye examination
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Saline 0.9%, volume will change to match that of dexmedetomidine based on participants' weight. 30 minutes before eye examination
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal administration of dexmedetomidine will be done using MAD Nasal atomization device (Teleflex Medical, 3015 Carrington Mill Blvd, Morrisville, NC 27560, USA). Administration will be given to both nares at a similar volume.
  Arms: Dexmedetomidine
Drug: Saline — Intranasal administration of saline 0.9% will be done using MAD Nasal atomization device (Teleflex Medical, 3015 Carrington Mill Blvd, Morrisville, NC 27560, USA). Administration will be given to both nares at a similar volume.
  Arms: Placebo

SUMMARY:
Background: Preterm infants undergo serial eye examinations during their hospital stay to monitor for the development of a specific disease termed "retinopathy of prematurity". While those examinations are known to cause significant pain and stress, the current standard of care (sucrose and local anesthesia) is not adequate in terms of alleviation of pain.

Purpose: The goal of this clinical trial is to test the effectiveness of dexmedetomidine for pain management in preterm infants undergoing routine eye examinations.

The main questions it aims to answer are:

* Does dexmedetomidine reduce the pain scores of preterm infants during and shortly after eye assessments in comparison to placebo (saline 0.9%).
* Does dexmedetomidine cause more adverse effects than placebo.

In this crossover study participants will receive either dexmedetomidine or saline 0.9% intranasally 30 minutes before the examination, on top of the current standard of care. The participants will be monitored closely for 5 hours to note differences in adverse effects. The researchers will use video monitoring to assess the pain scores using a standardized and validated scoring system.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 31 weeks post-menstrual age, or birth weight < 1500 grams
* Informed consent signed by one of the parents

Exclusion Criteria:

* Invasive ventilation at the time of the eye assessment
* Multiple congenital anomalies
* Chromosomal / genetic anomalies
* Infant received a sedative drug in last 5 days
* Eye examination for reasons other than retinopathy of prematurity screening
* Attending physician deemed the patient not stable enough

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The Premature Infant Pain Profile: Revised, at peak | PIPP-R score will be assessed 60 seconds after the insertion of the retractor
  The Premature Infant Pain Profile: Revised (PIPP-R) is a scoring system for pain and discomfort in preterm infants. The maximum attainable PIPP-R score is 21 for preterm infants <28 weeks GA and 18 for full-term infants. The higher the score, the greater the discomfort.
  Every participant will be assessed using video recordings which will start 5 minutes before the administration of oral sucrose 24% and will continue until 5 minutes after the removal of the eyelid retractor.
  The primary outcome will be the PIPP-R score one minute after the insertion of the retractor.

SECONDARY OUTCOMES:
The Premature Infant Pain Profile: Revised, 5 minutes | 5 minutes after the insertion of the retractor
  The Premature Infant Pain Profile: Revised (PIPP-R) is a scoring system for pain and discomfort in preterm infants. The maximum attainable PIPP-R score is 21 for preterm infants <28 weeks GA and 18 for full-term infants. The higher the score, the greater the discomfort.
  For this secondary outcome, PIPP-R score 5 minutes after the insertion of the retractor will be assessed.
The Premature Infant Pain Profile: Revised, at completion | 2 minutes after the removal the retractors
  The Premature Infant Pain Profile: Revised (PIPP-R) is a scoring system for pain and discomfort in preterm infants. The maximum attainable PIPP-R score is 21 for preterm infants <28 weeks GA and 18 for full-term infants. The higher the score, the greater the discomfort.
  For this secondary outcome, PIPP-R score 2 minutes after the after the removal the retractors will be assessed.
Apnea | From time 0 until 5 hours after the examination
  Number of apneas or desaturations < 90%
Bradycardia | From time 0 until 5 hours after the examination
  Number of bradycardias, defined as a drop of 20% from baseline heart rate
Heart rate | Assessed every hour from time 0 until 5 hours after the examination
  The average heart rate of the infant
Duration of examination | Up to 30 minutes
  The time between the insertion and the removal of the retractor
Percent of crying time | The duration of the video recording (up to 1 hour)
  The percent of time in which the participant cried during the video recording

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Be’er Ya‘aqov, Center, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wood EH, Chang EY, Beck K, Hadfield BR, Quinn AR, Harper CA 3rd. 80 Years of vision: preventing blindness from retinopathy of prematurity. J Perinatol. 2021 Jun;41(6):1216-1224. doi: 10.1038/s41372-021-01015-8. Epub 2021 Mar 5. PMID 33674712
- [Background] Chiang MF, Quinn GE, Fielder AR, Ostmo SR, Paul Chan RV, Berrocal A, Binenbaum G, Blair M, Peter Campbell J, Capone A Jr, Chen Y, Dai S, Ells A, Fleck BW, Good WV, Elizabeth Hartnett M, Holmstrom G, Kusaka S, Kychenthal A, Lepore D, Lorenz B, Martinez-Castellanos MA, Ozdek S, Ademola-Popoola D, Reynolds JD, Shah PK, Shapiro M, Stahl A, Toth C, Vinekar A, Visser L, Wallace DK, Wu WC, Zhao P, Zin A. International Classification of Retinopathy of Prematurity, Third Edition. Ophthalmology. 2021 Oct;128(10):e51-e68. doi: 10.1016/j.ophtha.2021.05.031. Epub 2021 Jul 8. PMID 34247850
- [Background] Nayak R, Nagaraj KN, Gururaj G. Prevention of Pain During Screening for Retinopathy of Prematurity: A Randomized Control Trial Comparing Breast Milk, 10% Dextrose and Sterile Water. Indian J Pediatr. 2020 May;87(5):353-358. doi: 10.1007/s12098-020-03182-6. Epub 2020 Jan 27. PMID 31989459
- [Background] Mitchell AJ, Green A, Jeffs DA, Roberson PK. Physiologic effects of retinopathy of prematurity screening examinations. Adv Neonatal Care. 2011 Aug;11(4):291-7. doi: 10.1097/ANC.0b013e318225a332. PMID 22123352
- [Background] Padhi TR, Sareen D, Pradhan L, Jalali S, Sutar S, Das T, Modi RR, Behera UC. Evaluation of retinopathy of prematurity screening in reverse Kangaroo Mother Care: a pilot study. Eye (Lond). 2015 Apr;29(4):505-8. doi: 10.1038/eye.2014.340. Epub 2015 Jan 23. PMID 25613847
- [Background] Valeri BO, Holsti L, Linhares MB. Neonatal pain and developmental outcomes in children born preterm: a systematic review. Clin J Pain. 2015 Apr;31(4):355-62. doi: 10.1097/AJP.0000000000000114. PMID 24866853
- [Background] Walker SM. Long-term effects of neonatal pain. Semin Fetal Neonatal Med. 2019 Aug;24(4):101005. doi: 10.1016/j.siny.2019.04.005. Epub 2019 Apr 5. PMID 30987942
- [Background] Nesargi SV, Nithyanandam S, Rao S, Nimbalkar S, Bhat S. Topical anesthesia or oral dextrose for the relief of pain in screening for retinopathy of prematurity: a randomized controlled double-blinded trial. J Trop Pediatr. 2015 Feb;61(1):20-4. doi: 10.1093/tropej/fmu058. Epub 2014 Nov 5. PMID 25376189
- [Background] Marsh VA, Young WO, Dunaway KK, Kissling GE, Carlos RQ, Jones SM, Shockley DH, Weaver NL, Ransom JL, Gal P. Efficacy of topical anesthetics to reduce pain in premature infants during eye examinations for retinopathy of prematurity. Ann Pharmacother. 2005 May;39(5):829-33. doi: 10.1345/aph.1E476. Epub 2005 Mar 29. PMID 15797982
- [Background] Disher T, Cameron C, Mitra S, Cathcart K, Campbell-Yeo M. Pain-Relieving Interventions for Retinopathy of Prematurity: A Meta-analysis. Pediatrics. 2018 Jul;142(1):e20180401. doi: 10.1542/peds.2018-0401. Epub 2018 Jun 1. PMID 29858451
- [Background] Dempsey E, McCreery K. Local anaesthetic eye drops for prevention of pain in preterm infants undergoing screening for retinopathy of prematurity. Cochrane Database Syst Rev. 2011 Sep 7;2011(9):CD007645. doi: 10.1002/14651858.CD007645.pub2. PMID 21901708
- [Background] Campbell-Yeo M, Benoit B. Use of morphine before retinopathy of prematurity examinations. Lancet. 2018 Dec 15;392(10164):2521-2523. doi: 10.1016/S0140-6736(18)32324-9. Epub 2018 Nov 30. No abstract available. PMID 30509742
- [Background] Alselaimy R, Al Tawil L, Abouammoh MA. Anesthesia in retinopathy of prematurity. Saudi J Ophthalmol. 2022 Oct 14;36(3):251-259. doi: 10.4103/sjopt.sjopt_229_21. eCollection 2022 Jul-Sep. PMID 36276254
- [Background] Hartley C, Moultrie F, Hoskin A, Green G, Monk V, Bell JL, King AR, Buckle M, van der Vaart M, Gursul D, Goksan S, Juszczak E, Norman JE, Rogers R, Patel C, Adams E, Slater R. Analgesic efficacy and safety of morphine in the Procedural Pain in Premature Infants (Poppi) study: randomised placebo-controlled trial. Lancet. 2018 Dec 15;392(10164):2595-2605. doi: 10.1016/S0140-6736(18)31813-0. Epub 2018 Nov 30. PMID 30509743
- [Background] Sindhur M, Balasubramanian H, Srinivasan L, Kabra NS, Agashe P, Doshi A. Intranasal fentanyl for pain management during screening for retinopathy of prematurity in preterm infants: a randomized controlled trial. J Perinatol. 2020 Jun;40(6):881-887. doi: 10.1038/s41372-020-0608-2. Epub 2020 Feb 13. PMID 32054982
- [Background] McDonald D, Palsgraf H, Shah P. Dexmedetomidine - An emerging option for sedation in neonatal patients. J Perinatol. 2022 Jul;42(7):845-855. doi: 10.1038/s41372-022-01351-3. Epub 2022 Feb 23. PMID 35197548
- [Background] O'Mara K, Gal P, Wimmer J, Ransom JL, Carlos RQ, Dimaguila MA, Davanzo CC, Smith M. Dexmedetomidine versus standard therapy with fentanyl for sedation in mechanically ventilated premature neonates. J Pediatr Pharmacol Ther. 2012 Jul;17(3):252-62. doi: 10.5863/1551-6776-17.3.252. PMID 23258968
- [Background] Laudenbach V, Mantz J, Lagercrantz H, Desmonts JM, Evrard P, Gressens P. Effects of alpha(2)-adrenoceptor agonists on perinatal excitotoxic brain injury: comparison of clonidine and dexmedetomidine. Anesthesiology. 2002 Jan;96(1):134-41. doi: 10.1097/00000542-200201000-00026. PMID 11753013
- [Background] Lewis J, Bailey CR. Intranasal dexmedetomidine for sedation in children; a review. J Perioper Pract. 2020 Jun;30(6):170-175. doi: 10.1177/1750458919854885. Epub 2019 Jun 27. PMID 31246159
- [Background] Bua J, Massaro M, Cossovel F, Monasta L, Brovedani P, Cozzi G, Barbi E, Demarini S, Travan L. Intranasal dexmedetomidine, as midazolam-sparing drug, for MRI in preterm neonates. Paediatr Anaesth. 2018 Aug;28(8):747-748. doi: 10.1111/pan.13454. No abstract available. PMID 30144232
- [Background] Yuen VM, Hui TW, Irwin MG, Yao TJ, Wong GL, Yuen MK. Optimal timing for the administration of intranasal dexmedetomidine for premedication in children. Anaesthesia. 2010 Sep;65(9):922-9. doi: 10.1111/j.1365-2044.2010.06453.x. PMID 20645951
- [Background] Stevens BJ, Gibbins S, Yamada J, Dionne K, Lee G, Johnston C, Taddio A. The premature infant pain profile-revised (PIPP-R): initial validation and feasibility. Clin J Pain. 2014 Mar;30(3):238-43. doi: 10.1097/AJP.0b013e3182906aed. PMID 24503979
- [Background] Slater R, Hartley C, Moultrie F, Adams E, Juszczak E, Rogers R, Norman JE, Patel C, Stanbury K, Hoskin A, Green G; Poppi Trial Team. A blinded randomised placebo-controlled trial investigating the efficacy of morphine analgesia for procedural pain in infants: Trial protocol. Wellcome Open Res. 2016 Nov 15;1:7. doi: 10.12688/wellcomeopenres.10005.2. PMID 28066825